CLINICAL TRIAL: NCT02347956
Title: The Safety and Feasibility of Reduced Port Robotic Distal Gastrectomy Using Single-site for Surgical Treatment of Early Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0864
Record Dates: First submitted 2015-01-20; First posted 2015-01-28 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Gastric Cancer
Keywords: robot surgery; reduced port; single-site; safety; feasibility
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reduced port group (Experimental)
  Interventions: Procedure: Reduced port robotic distal gastrectomy

INTERVENTIONS:
Procedure: Reduced port robotic distal gastrectomy

SUMMARY:
Gastric cancer is one of the most common malignancy worldwide. Surgical resection of the tumor is the only curative treatment for gastric cancer. However, surgical procedure accompanies postoperative pain and prolonged hospitalization. To lessen the surgical trauma and stress, minimally invasive surgery were introduced. Laparoscopic gastrectomy was accepted as safe and effective alternative to open gastrectomy. Furthermore, reduced port and single port laparoscopic gastrectomy are considered to minimize the surgical trauma during gastrectomy. However, limitations of laparoscopic approach using reduced port includes unergonomic posture of surgeon, physiologic tremor and collision of instruments. To overcome these limitations, robot surgery using novel single-site technology enabled surgeons to perform the surgical procedure reducing the number of trocar from three to one for insertion of scope and two robotic arms. Previously, successful application of single-site technology for cholecystectomy and hysterectomy were reported. The aim of this study is to validate the safety and feasibility of reduced port robotic distal gastrectomy using single-site technology for the surgical treatment of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. A resectable, tissue confirmed adenocarcinoma of the stomach
2. Early gastric cancer curable by distal gastrectomy
3. AGE: 20-70
4. ECOG: 0-1
5. ASA score 1-3
6. A patient who signed the informed consent

Exclusion Criteria:

1. Advanced lesion with metastatic cancer
2. lesion which is curable by EMR or ESD
3. Previous major abdominal surgery
4. Complicated gastric cancer (obstruction or perforation)
5. History with other primary tumor within 5 year
6. Active other primary tumor
7. Vulnerable subjects (pregnant women, illiterate)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
morbidity | 30 days

SECONDARY OUTCOMES:
mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Jeong O, Park YK. Clinicopathological features and surgical treatment of gastric cancer in South Korea: the results of 2009 nationwide survey on surgically treated gastric cancer patients. J Gastric Cancer. 2011 Jun;11(2):69-77. doi: 10.5230/jgc.2011.11.2.69. Epub 2011 Jun 30. PMID 22076206
- [Background] Kim HH, Hyung WJ, Cho GS, Kim MC, Han SU, Kim W, Ryu SW, Lee HJ, Song KY. Morbidity and mortality of laparoscopic gastrectomy versus open gastrectomy for gastric cancer: an interim report--a phase III multicenter, prospective, randomized Trial (KLASS Trial). Ann Surg. 2010 Mar;251(3):417-20. doi: 10.1097/SLA.0b013e3181cc8f6b. PMID 20160637
- [Background] Kim YM, Baek SE, Lim JS, Hyung WJ. Clinical application of image-enhanced minimally invasive robotic surgery for gastric cancer: a prospective observational study. J Gastrointest Surg. 2013 Feb;17(2):304-12. doi: 10.1007/s11605-012-2094-0. Epub 2012 Dec 1. PMID 23207683
- [Background] Kitano S, Iso Y, Moriyama M, Sugimachi K. Laparoscopy-assisted Billroth I gastrectomy. Surg Laparosc Endosc. 1994 Apr;4(2):146-8. PMID 8180768
- [Background] Lee JH, Kim KM, Cheong JH, Noh SH. Current management and future strategies of gastric cancer. Yonsei Med J. 2012 Mar;53(2):248-57. doi: 10.3349/ymj.2012.53.2.248. PMID 22318810
- [Background] Pietrabissa A, Sbrana F, Morelli L, Badessi F, Pugliese L, Vinci A, Klersy C, Spinoglio G. Overcoming the challenges of single-incision cholecystectomy with robotic single-site technology. Arch Surg. 2012 Aug;147(8):709-14. doi: 10.1001/archsurg.2012.508. PMID 22508669
- [Background] Tokunaga M, Sugisawa N, Kondo J, Tanizawa Y, Bando E, Kawamura T, Terashima M. Early phase II study of robot-assisted distal gastrectomy with nodal dissection for clinical stage IA gastric cancer. Gastric Cancer. 2014;17(3):542-7. doi: 10.1007/s10120-013-0293-3. Epub 2013 Sep 5. PMID 24005955
- [Background] Vizza E, Corrado G, Mancini E, Baiocco E, Patrizi L, Fabrizi L, Colantonio L, Cimino M, Sindico S, Forastiere E. Robotic single-site hysterectomy in low risk endometrial cancer: a pilot study. Ann Surg Oncol. 2013 Aug;20(8):2759-64. doi: 10.1245/s10434-013-2922-9. Epub 2013 Mar 7. PMID 23468046
- [Background] Zeng YK, Yang ZL, Peng JS, Lin HS, Cai L. Laparoscopy-assisted versus open distal gastrectomy for early gastric cancer: evidence from randomized and nonrandomized clinical trials. Ann Surg. 2012 Jul;256(1):39-52. doi: 10.1097/SLA.0b013e3182583e2e. PMID 22664559